CLINICAL TRIAL: NCT03081117
Title: Clinical Trial of Intranasal Insulin for the Treatment of HIV-associated Neurocognitive Disorder (HAND)
Brief Title: Intranasal Insulin for the Treatment of HAND
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: On 3/15/2020 study visits were suspended due to COVID-19 pandemic. With safety concerns surrounding COVID-19 and difficulty recruiting, the investigators decided to close enrollment 10/16/2020 after interim data were reviewed by the DSMB and NIH.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00108564
Record Dates: First submitted 2017-03-09; First posted 2017-03-16 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: HIV Dementia; HIV-Associated Cognitive Motor Complex
Keywords: HIV-Associated Neurocognitive Disorder (HAND); Intranasal
MeSH Terms: conditions — AIDS Dementia Complex | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin, intranasal (Experimental): Regular insulin, 20 IU intranasal twice a day for 24 weeks; 0.2 mL per dose
  Interventions: Drug: Insulin, intranasal
- Placebo, intranasal (Placebo Comparator): Saline solution (placebo), intranasal twice a day for 24 weeks; 0.2 mL per dose
  Interventions: Drug: Placebo, intranasal

INTERVENTIONS:
Drug: Insulin, intranasal — Regular insulin administered by specialized, non-commercial intranasal drug delivery device
  Other Names: Novolin R
  Arms: Insulin, intranasal
Drug: Placebo, intranasal — Saline solution administered by specialized, non-commercial intranasal drug delivery device
  Arms: Placebo, intranasal

SUMMARY:
Infection with HIV (the virus that causes AIDS) can lead to problems with brain function, such as memory, concentration, judgment, and the speed or control of hands and legs. Neurologists have called this condition HIV-associated neurocognitive disorder (HAND). This research is being done to see if insulin taken through the nose as a spray (intranasal insulin) can help people with HIV who are having problems with memory and brain function, or HAND.

Participants will be given either insulin or placebo. A placebo is an inactive substance that looks like the study drug, but does not contain study drug. For this research study, the placebo will be a clear, saline-based liquid spray that looks like the insulin spray but has no insulin. Participants will not be told whether they receive insulin or placebo during the study.

All participants will take the intranasal spray twice a day, about 30 minutes after a meal. Participants will use a specialized intranasal drug administration device. The total daily dose of insulin is 40 IU split between 20 IU in the morning and 20 IU in the evening. Participants will take the intranasal spray for 24 weeks.

The researchers will record symptoms and side effects during the study. Procedures include neurocognitive testing of memory and brain function, two optional lumbar punctures ("spinal taps"), two MRI brain scans, monthly blood draws, and clinical assessments.

DETAILED DESCRIPTION:
HIV-associated neurocognitive disorders (HAND) are characterized by disabling cognitive, behavioral, and motor dysfunction and can occur in individuals with HIV even while taking combination antiretroviral therapy (ART). The mechanisms for these residual impairments are not fully understood, but appear to involve poor penetrance of ART drugs into the central nervous system (CNS) and the resulting brain sanctuary for inadequately suppressed HIV infection with associated sustained inflammation. Adjunctive therapies with targeted neuroprotective agents are critically needed for the treatment of HAND. Insulin is involved in multiple CNS functions including food intake, metabolism, learning, and memory. Insulin has neuroprotective properties demonstrated in cell culture experiments and in vivo models, which provide strong evidence for its use as a therapeutic agent to treat HAND.

Insulin modifying therapy (IMT) includes intranasal insulin administered by a novel nasal drug delivery device. IMT may play important roles in neuronal plasticity and survival by protecting hippocampal neurons against oxidative stress and apoptotic cell death induced by glutamate neurotoxicity. Previous studies support the proposed early phase trial of IMT as a novel therapeutic agent for HAND.

This double-blinded placebo-controlled clinical trial evaluates safety of intranasal insulin at the daily dose of 40 IU and will provide initial data for assessing safety and efficacy. The protocol measures safety by incidence and frequency of adverse events. Clinical effects of IMT over the 24-week trial period are measured by change in neurocognitive and functional testing results, as well as several novel radiological and cerebrospinal fluid (CSF) surrogate markers. Outcomes from these studies could have important implications for the design of future studies with IMT and other neuroprotective compounds for HAND.

ELIGIBILITY:
Inclusion Criteria:

* Must have HIV,
* Capable of providing informed consent,
* Between the ages of 18-69 years,
* Evidence of problems with memory, speed, and brain function,
* Same HIV medications for at least 6 months (180 days) prior to study entry, with no plans to change the medications over the study period,
* The following blood lab values within 2 weeks prior to study entry: hemoglobin > 8.9 g/dl, absolute neutrophil count > 500 cells/mm3, platelet count > 50,000 cells/mm3, alanine aminotransferase (ALT) < 2.5 X upper limit of normal, alkaline phosphatase < 3 X upper limit of normal, serum creatinine ≤ 2 X upper limit of normal,
* Negative pregnancy test (for women who could become pregnant),
* Able and willing to use an intranasal device for taking the study drug without complications (e.g., no history of traumatic obstruction to nasal passage, chronic sinus infections, severe and symptomatic seasonal allergies, etc.),
* Currently suppressed blood HIV viral load (undetectable or <400 copies/mL).

Exclusion Criteria:

* Current or past opportunistic infection of the brain,
* History or current clinical evidence of schizophrenia,
* History of chronic neurological disorder, such as multiple sclerosis or uncontrolled epilepsy,
* Active symptomatic AIDS defining opportunistic infection within 30 days prior to study entry,
* History of an uncontrolled medical or psychiatric illness which in the opinion of the investigators would constitute a safety risk for patients or interfere with the ability of a participant to complete the study,
* History of diabetes or treatment with insulin or an oral hypoglycemic agent,
* Amylase/lipase elevation (≥ 2 X upper limit of normal) within 14 days prior to starting study drug,
* Detectable plasma HIV RNA test ≥400 copies/mL within 6 months prior to baseline/randomization,
* History of any endocrine related cancer, including any thyroid tumor,
* Current use of cocaine, heroin, or methamphetamine. Current use will be defined and determined by any evidence of such use within the two years (730 days) prior to study enrollment; evidence includes but is not limited to urine drug toxicology testing by the study team at screening and pre-entry visits,
* Presence of other conditions that significantly affect and complicate performance on neurocognitive tests (such as, learning disabilities, history of severe alcohol abuse, head injury with trauma to the brain and loss of consciousness >30 minutes).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah Rubin, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Institute for Clinical and Translational Research, Adult Outpatient Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Started | 10 | 11
Primary Outcome 1 (SAE) (Participants who received at least 12 weeks of follow-up monitoring to collect serious adverse event (SAE) data.) | 10 | 11
Secondary Measures Collected at Week 24 (Participants with at least secondary measures collected at 24 weeks.) | 8 | 9
Completed (ITT): Primary Outcome 2 (GDS) (Participants who completed neurocognitive test measures with valid Global Deficit Score (GDS) at 24 weeks.) | 7 | 9
Completed (Valid primary outcome measures and compliance with study intervention >66% (16 Weeks).) | 6 | 8
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin, Intranasal | Placebo, Intranasal | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  years
    Enrolled | 58.5 [55 to 61] | 58 [56 to 62] | 58 [56 to 61]
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 57 [54.5 to 61.5] | 58 [56 to 62] | 57.5 [55 to 62.25]
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 56 [54.25 to 57.75] | 57.5 [55.75 to 59.25] | 57 [55 to 59.5]
Age, Customized [Count of Participants; unit: Participants] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  Participants
    Enrolled: 30-39 | 1 | 0 | 1
    Enrolled: 40-49 | 0 | 1 | 1
    Enrolled: 50-59 | 5 | 5 | 10
    Enrolled: 60-69 | 4 | 5 | 9
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT): 30-39 | 1 | 0 | 1
    Completed Trial (ITT): 40-49 | 0 | 1 | 1
    Completed Trial (ITT): 50-59 | 4 | 5 | 9
    Completed Trial (ITT): 60-69 | 2 | 3 | 5
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol): 30-39 | 1 | 0 | 1
    Completed Trial (Per Protocol): 40-49 | 0 | 1 | 1
    Completed Trial (Per Protocol): 50-59 | 4 | 5 | 9
    Completed Trial (Per Protocol): 60-69 | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  Participants
    Enrolled: Female | 3 | 5 | 8
    Enrolled: Male | 7 | 6 | 13
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT): Female | 3 | 4 | 7
    Completed Trial (ITT): Male | 4 | 5 | 9
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol): Female | 3 | 3 | 6
    Completed Trial (Per Protocol): Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
Education, Continuous [Mean (Standard Deviation); unit: years] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  years
    Enrolled | 12.70 (2.06) | 12.09 (1.87) | 12.38 (1.94)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 12.86 (2.34) | 12.33 (1.94) | 12.56 (2.06)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 12.33 (2.07) | 12.50 (2.00) | 12.43 (1.95)
Education, Categorical [Count of Participants; unit: Participants] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  Participants
    Enrolled: 9th to 11th Grade | 2 | 3 | 5
    Enrolled: High School Diploma | 4 | 6 | 10
    Enrolled: Some College or Associates Degree | 3 | 1 | 4
    Enrolled: College Degree | 1 | 1 | 2
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT): 9th to 11th Grade | 1 | 2 | 3
    Completed Trial (ITT): High School Diploma | 3 | 5 | 8
    Completed Trial (ITT): Some College or Associates Degree | 2 | 1 | 3
    Completed Trial (ITT): College Degree | 1 | 1 | 2
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol): 9th to 11th Grade | 1 | 1 | 2
    Completed Trial (Per Protocol): High School Diploma | 3 | 5 | 8
    Completed Trial (Per Protocol): Some College or Associates Degree | 2 | 1 | 3
    Completed Trial (Per Protocol): College Degree | 0 | 1 | 1
Global Deficit Score (GDS), Baseline [Mean (Standard Deviation); unit: units on a scale] — GDS is a composite score of neurocognitive test performance comprised of 14 data points from 9 tests (Hopkins Verbal Learning, Rey Complex Figure, WAIS symbol-digit, grooved pegboard, CalCAP, Trail-making, Stroop Color Interference, timed gait, and FAS verbal fluency). Raw scores were transformed to t-scores using age/education stratified norms, assigned discrete values 0 to 5 (t-score categorization > or =40 is 0, 35.00 to 39.99 =1, 30.00 to 34.99 =2, 25.00 to 29.99 =3, 20.00 to 24.99 =4, and <20 =5) and then averaged. Higher GDS is a worse outcome (0 = no deficits and 5 = maximum deficits). Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  units on a scale
    Enrolled | 1.37 (0.74) | 0.85 (0.57) | 1.10 (0.70)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 1.31 (0.56) | 0.75 (0.47) | 1.00 (0.57)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 1.22 (0.55) | 0.77 (0.50) | 0.97 (0.55)
Beck Depression Inventory II [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory II is a standard 21-item paper questionnaire in which participants self-rated signs and symptoms of depression over the preceding 2 weeks. Each item was scored 0, 1, 2, or 3, and then added up for a total score (test range: 0 - 63) with higher numbers indicating greater severity of depressive symptoms. Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  units on a scale
    Enrolled | 10.10 (7.95) | 5.55 (4.08) | 7.71 (6.50)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 9.14 (7.84) | 5.44 (4.56) | 7.06 (6.27)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 10.67 (7.37) | 5.88 (4.67) | 7.93 (6.22)
Beck Depression Inventory II [Median (Inter-Quartile Range); unit: units on a scale] — The Beck Depression Inventory II is a standard 21-item paper questionnaire in which participants self-rated signs and symptoms of depression over the preceding 2 weeks. Each item was scored 0, 1, 2, or 3, and then added up for a total score (test range: 0 - 63) with higher numbers indicating greater severity of depressive symptoms. Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  units on a scale
    Enrolled | 11.0 [3.50 to 15.50] | 6.0 [2.00 to 7.50] | 6.0 [2.00 to 13.00]
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 13.0 [1.50 to 15.00] | 4.0 [2.00 to 9.00] | 5.0 [1.75 to 13.00]
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 13.5 [5.50 to 15.50] | 5.0 [1.75 to 9.50] | 7.5 [2.25 to 13.00]
Estimated IQ, Hopkins Adult Reading Test [Mean (Standard Deviation); unit: units on a scale] — The Hopkins Adult Reading Test (HART) is a standard 35 item word list that the participant reads while the tester assesses his/her pronunciation of each word. One point is awarded for each correct pronunciation (raw score range 0-35). The number correct is then transformed to a standard score based on age/education/sex/race matched normative data with the mean set to 100 and standard deviation of 15 (range defined valid between 73 and 131). Higher scores indicate greater word recognition. It serves as an estimated measure of premorbid abilities (i.e. Intelligence Quotient). Population: Two participants did not perform the Hopkins Adult Reading Test at baseline. Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  units on a scale
    Enrolled: number analyzed (Participants) | 8 | 11 | 19
    Enrolled | 97.13 (6.64) | 96.00 (11.54) | 96.47 (9.56)
    Completed Trial (ITT): number analyzed (Participants) | 6 | 9 | 15
    Completed Trial (ITT) | 98.67 (6.50) | 97.67 (12.22) | 98.07 (10.03)
    Completed Trial (Per Protocol): number analyzed (Participants) | 5 | 8 | 13
    Completed Trial (Per Protocol) | 98.80 (7.26) | 98.63 (12.69) | 98.69 (10.56)
Hopkins Verbal Learning Test, Total (Trials 1-3) [Mean (Standard Deviation); unit: z-score] — The total sum of correct words immediately recalled over three trials. The raw scores were transformed to Z-scores based on an age-matched reference population. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of the reference population with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate a greater verbal learning score (better outcome). Z-scores under -3.5 were limited to -3.5. Population: Measure Analysis Population Description: Enrolled: All participants started on study intervention.
  Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  z-score
    Enrolled | -1.41 (1.00) | -0.96 (0.82) | -1.18 (0.92)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | -1.56 (1.15) | -1.01 (0.91) | -1.25 (1.02)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | -1.34 (1.09) | -0.84 (0.80) | -1.06 (0.93)
Hopkins Verbal Learning Test, Delayed Recall [Mean (Standard Deviation); unit: z-score] — Total words recalled after 20 minute delay. The raw scores were transformed to Z-scores based on an age-matched reference population. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of the reference population with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate a greater verbal learning score (better outcome). Z-scores under -3.5 were limited to -3.5. Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  z-score
    Enrolled | -2.00 (1.50) | -1.20 (0.98) | -1.58 (1.29)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | -2.10 (1.74) | -0.93 (0.67) | -1.44 (1.34)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | -1.89 (1.80) | -0.88 (0.70) | -1.31 (1.33)
Rey Complex Figure Test, Copy [Mean (Standard Deviation); unit: z-score] — Standard Rey Complex Figure scoring applied to assess ability to copy the test figure (range 0-36). The raw scores were transformed to Z-scores based on age-matched reference population data. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of the reference population with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate a greater visual-spatial reconstruction score (better outcome). Z-scores under -3.5 were limited to -3.5. Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  z-score
    Enrolled | -2.20 (1.32) | -1.15 (1.14) | -1.65 (1.31)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | -2.39 (1.25) | -1.12 (1.27) | -1.67 (1.38)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | -2.20 (1.26) | -0.91 (1.20) | -1.47 (1.35)
Rey Complex Figure Test, Delayed Recall [Mean (Standard Deviation); unit: z-score] — Standard Rey Complex Figure scoring applied to assess ability to recall the test figure after 20 minutes (range 0-36). The raw scores were transformed to Z-scores based on age-matched reference population data. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of the reference population with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate a greater visual-spatial recall score (better outcome). Z-scores under -3.5 were limited to -3.5. Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  z-score
    Enrolled | -0.87 (0.95) | -0.46 (0.91) | -0.65 (0.93)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | -0.63 (0.92) | -0.27 (0.90) | -0.43 (0.90)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | -0.46 (0.87) | -0.19 (0.93) | -0.31 (0.88)
Trail Making Test, Part A [Mean (Standard Deviation); unit: z-score] — Time to complete Trail Making Test Part A. The raw scores (measured in seconds) were transformed to directionally inverted Z-scores based on age/education/sex-matched reference population data. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of the reference population. The inverted Z-scores produce negative numbers when times are higher than the mean and positive values when times are lower. Higher Z-scores indicate a greater motor speed (better outcome). Z-scores under -3.5 were limited to -3.5. Population: Measure Analysis Population Description: Enrolled: All participants started on study intervention.
  Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  z-score
    Enrolled | -0.94 (0.61) | -0.02 (0.72) | -0.46 (0.81)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | -0.91 (0.48) | 0.02 (0.76) | -0.39 (0.79)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | -0.88 (0.52) | -0.16 (0.56) | -0.47 (0.64)
Trail Making Test, Part B [Mean (Standard Deviation); unit: z-score] — Time to complete Trail Making Test Part B. The raw scores (measured in seconds) were transformed to directionally inverted Z-scores based on age/education/sex-matched reference population data. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of the reference population. The inverted Z-scores produce negative numbers when times are higher than the mean and positive values when times are lower. Higher Z-scores indicate a greater motor speed (better outcome). Z-scores under -3.5 were limited to -3.5. Population: Two participants were unable to complete test in the allotted time. Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  z-score
    Enrolled: number analyzed (Participants) | 9 | 10 | 19
    Enrolled | -0.76 (0.59) | -0.23 (0.64) | -0.48 (0.66)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | -0.66 (0.62) | -0.14 (0.62) | -0.37 (0.65)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | -0.63 (0.67) | -0.13 (0.66) | -0.34 (0.69)
Grooved Pegboard Test, Dominant Hand [Mean (Standard Deviation); unit: z-score] — Time to complete grooved pegboard task with dominant hand. The raw scores (measured in seconds) were transformed to directionally inverted Z-scores based on age/education/sex-matched reference population data. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of the reference population. The inverted Z-scores produce negative numbers when times are higher than the mean and positive values when times are lower. Higher Z-scores indicate a greater motor speed (better outcome). Z-scores under -3.5 were limited to -3.5. Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  z-score
    Enrolled | -0.83 (1.09) | -0.78 (0.49) | -0.80 (0.81)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | -0.74 (0.97) | -0.83 (0.50) | -0.79 (0.72)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | -0.68 (1.05) | -0.90 (0.50) | -0.81 (0.75)
Grooved Pegboard Test, Non-Dominant Hand [Mean (Standard Deviation); unit: z-score] — Time to complete grooved pegboard task with non-dominant hand. The raw scores (measured in seconds) were transformed to directionally inverted Z-scores based on age/education/sex-matched reference population data. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of the reference population. The inverted Z-scores produce negative numbers when times are higher than the mean and positive values when times are lower. Higher Z-scores indicate a greater motor speed (better outcome). Z-scores under -3.5 were limited to -3.5. Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  z-score
    Enrolled | -1.42 (1.07) | -0.35 (1.46) | -0.86 (1.37)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | -1.41 (1.05) | -0.38 (1.56) | -0.83 (1.42)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | -1.27 (1.07) | -0.76 (1.11) | -0.98 (1.08)
CD4, Absolute Count [Mean (Standard Deviation); unit: cells per cubic mm] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  cells per cubic mm
    Enrolled | 616.80 (170.18) | 598.55 (290.86) | 607.24 (235.41)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 538.86 (127.73) | 527.78 (176.30) | 532.63 (152.10)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 518.17 (126.42) | 514.63 (183.69) | 516.14 (155.95)
HIV Viral Load, Plasma [Count of Participants; unit: Participants] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  Participants
    Enrolled: Undetectable (<20 copies/mL) | 5 | 9 | 14
    Enrolled: Low Detectable (20-49 copies/mL) | 5 | 1 | 6
    Enrolled: Low Detectable (50-99 copies/mL) | 0 | 1 | 1
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT): Undetectable (<20 copies/mL) | 3 | 7 | 10
    Completed Trial (ITT): Low Detectable (20-49 copies/mL) | 4 | 1 | 5
    Completed Trial (ITT): Low Detectable (50-99 copies/mL) | 0 | 1 | 1
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol): Undetectable (<20 copies/mL) | 2 | 6 | 8
    Completed Trial (Per Protocol): Low Detectable (20-49 copies/mL) | 4 | 1 | 5
    Completed Trial (Per Protocol): Low Detectable (50-99 copies/mL) | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  kg/m^2
    Enrolled | 31.33 (8.38) | 31.45 (6.83) | 31.40 (7.41)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 31.13 (9.60) | 30.24 (5.73) | 30.63 (7.39)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 32.38 (9.86) | 30.44 (6.10) | 31.27 (7.64)
Glucose, Fasting Blood [Mean (Standard Deviation); unit: mg/dL] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  mg/dL
    Enrolled | 101.50 (11.68) | 93.55 (11.11) | 97.33 (11.82)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 101.86 (13.69) | 93.33 (12.35) | 97.06 (13.24)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 101.83 (15.00) | 95.63 (10.97) | 98.29 (12.71)
Insulin, Fasting Serum [Mean (Standard Deviation); unit: mcU/mL] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  mcU/mL
    Enrolled | 29.38 (31.93) | 42.66 (82.28) | 36.34 (62.37)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 25.23 (38.18) | 19.30 (17.43) | 21.89 (27.47)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 28.77 (40.55) | 19.83 (18.56) | 23.66 (28.96)
Amylase, Blood [Mean (Standard Deviation); unit: U/L] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  U/L
    Enrolled | 89.00 (30.32) | 78.73 (27.53) | 83.62 (28.64)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 89.14 (35.43) | 80.11 (30.51) | 84.06 (31.93)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 88.83 (38.80) | 82.50 (31.70) | 85.21 (33.63)
Lipase, Blood [Mean (Standard Deviation); unit: U/L] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  U/L
    Enrolled | 25.70 (9.70) | 28.55 (12.68) | 27.19 (11.17)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 22.14 (8.53) | 27.44 (13.90) | 25.13 (11.81)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 23.67 (8.24) | 26.13 (14.25) | 25.07 (11.70)
Thyroid Stimulating Hormone [Mean (Standard Deviation); unit: u[IU]/mL] — Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  u[IU]/mL
    Enrolled | 1.67 (0.34) | 1.50 (0.78) | 1.58 (0.60)
    Completed Trial (ITT): number analyzed (Participants) | 7 | 9 | 16
    Completed Trial (ITT) | 1.52 (0.19) | 1.69 (0.73) | 1.62 (0.55)
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8 | 14
    Completed Trial (Per Protocol) | 1.50 (0.20) | 1.72 (0.77) | 1.63 (0.59)
Vitamin B12, Blood [Median (Inter-Quartile Range); unit: pg/mL] — Population: Two participants did not have baseline vitamin B12 levels tested. Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
  pg/mL
    Enrolled: number analyzed (Participants) | 10 | 9 | 19
    Enrolled | 390.5 [291.50 to 573.00] | 448.0 [417.00 to 540.00] | 442.0 [323.00 to 565.50]
    Completed Trial (ITT): number analyzed (Participants) | 7 | 8 | 15
    Completed Trial (ITT) | 397.0 [332.50 to 555.00] | 461.0 [393.50 to 645.25] | 448.0 [353.50 to 565.50]
    Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 7 | 13
    Completed Trial (Per Protocol) | 390.5 [306.75 to 488.50] | 474.0 [385.50 to 750.50] | 448.0 [323.00 to 540.00]

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Event Frequency
Description: Number of documented serious adverse events per participant, mean
Time Frame: Total during 24-week trial
Population: Enrolled: All participants started on study intervention. Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
Measure: Mean (Standard Deviation); unit: Number of SAEs/participant
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 10 | 11
Number of SAEs/participant
  Enrolled | 0.30 (0.67) | 0.18 (0.40)
  Completed Trial (ITT): number analyzed (Participants) | 7 | 9
  Completed Trial (ITT) | 0.14 (0.38) | 0.22 (0.44)
  Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8
  Completed Trial (Per Protocol) | 0.00 (0.00) | 0.25 (0.46)

2. Primary Outcome: Serious Adverse Event Frequency, Participant Count
Description: Number participants with at least one documented serious adverse event, count
Time Frame: Total during 24-week trial
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 10 | 11
Participants
  Enrolled | 2 | 2
  Completed Trial (ITT): number analyzed (Participants) | 7 | 9
  Completed Trial (ITT) | 1 | 2
  Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8
  Completed Trial (Per Protocol) | 0 | 2
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; Analysis of Enrolled group; Test type: Superiority; p = 0.669, Fisher Exact

3. Primary Outcome: Neurocognitive Performance: Global Deficit Score (GDS), Week 24 Visit Score Minus Baseline Score
Description: Change in GDS, measured at two time points, baseline and Week 24 visits. GDS is a composite score based on neurocognitive test performance. The 14 data points that comprise the GDS include Hopkins Verbal Learning Test (trials 1-3 total score and delayed recall), Rey Complex Figure Test (copy and delayed recall), WAIS symbol-digit test, grooved pegboard (dominant and non-dominant), CalCAP (Choice reaction time and Sequential reaction time), Trail-making Test (Parts A and B), Stroop Color Interference Test (trial 3), timed gait (3 trials average), and verbal fluency (FAS). Raw scores were transformed to t-scores using age/education stratified normative data, then assigned a discrete value from 0 to 5 using the following t-score categorization: > or = 40 is '0', 35.00 to 39.99 is '1', 30.00 to 34.99 is '2', 25.00 to 29.99 is '3', 20.00 to 24.99 is '4', and <20 is '5'. The 14 individual scores were then averaged. A higher GDS is a worse outcome (0 = no deficits and 5 = maximum deficits).
Time Frame: Difference between baseline and week 24 visits
Population: Completed Trial (ITT): All participants with both primary outcome measures at 24 weeks.
  Completed Trial (Per Protocol): Participants with both primary outcome measures at 24 weeks and who demonstrated greater than 16 weeks adherence to the study intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 7 | 9
units on a scale
  Completed Trial (ITT) | -0.1614 (0.3810) | 0.2300 (0.2981)
  Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8
  Completed Trial (Per Protocol) | -0.2383 (0.3529) | 0.2763 (0.2820)
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; Analysis for Intent-to-Treat group; Test type: Superiority; p = 0.0366, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees of freedom = 14; Mean Difference (Net) = -0.3914
Statistical Analysis 2: Comparison: Insulin, Intranasal vs Placebo, Intranasal; Analysis for Per Protocol group; Test type: Superiority; p = 0.0103, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees of freedom = 12; Mean Difference (Net) = -0.5146

4. Secondary Outcome: Neurocognitive Performance: NPZ-8 Score, Week 24 Visit Score Minus Baseline Score
Description: NPZ-8 score at 24 weeks minus baseline NPZ-8 score: The NPZ-8 is an average of 8 individual Z-scores, where higher values indicate greater neurocognitive performance (better outcome). The NPZ-8 represents the number of standard deviations an individual's performance is away from the mean (Z-score = 0) of age and education matched reference populations where performance worse than the mean had negative Z-scores (i.e. Z-scores were inverted for tests scored on speed). The NPZ-8 average is comprised of 8 data points from 6 tests: timed gait, WAIS symbol-digit, grooved pegboard dominant & non-dominant, CalCAP Choice & Sequential reaction times, and the Trail-making Test parts A & B. Raw scores were transformed to Z-scores for each test and then averaged to calculate the NPZ-8 score at each visit (Z-scores +/-3.5 standard deviations from mean limited to +/-3.5). Positive change in NPZ-8 from baseline to Week 24 indicated improved performance and negative change indicated worse performance.
Time Frame: Difference between baseline and week 24 visits
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 7 | 9
z-score
  Completed Trial (ITT) | -0.09 (0.39) | -0.01 (0.57)
  Completed Trial (Per Protocol): number analyzed (Participants) | 6 | 8
  Completed Trial (Per Protocol) | -0.07 (0.42) | -0.02 (0.60)

5. Secondary Outcome: CSF Biomarkers, Week 24 Visit Value Minus Baseline Value
Description: Changes in cerebrospinal fluid (CSF) concentrations of ceramide, sphingomyelin, citrate, neurofilament protein; brain-derived neurotrophic factor (BDNF), protein carbonyl, Aβ-42
Time Frame: Between baseline and week 24 visits
Population: Baseline and Week 24 CSF samples were collected from only 4 participants. CSF biomarker assays were not performed because the target number of 36 evaluable patients was not reached, and we had insufficient power to detect a true difference in change per the statistical analysis plan.
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Neuroimaging Markers: SV-MRS, Myoinositol, Basal Ganglia, Week 24 Visit Value Minus Baseline Value
Description: Single voxel-magnetic resonance spectroscopy (SV-MRS) myoinositol in the basal ganglia. Results were reported as concentrations measured in approximated mmol/L (institutional units).
Time Frame: Changes between baseline and week 24 visits
Population: MRS was performed at both baseline and 24 Weeks on 16 participants (Pts). However, one had invalid basal ganglia MRS results at Week 24, another is missing all Week 24 MRS results due to technical error in data collection.
  Available MRS (data for outcome measure): 14 Pts. (Note: one of the Pts did not complete trial, two were Intent-to-Treat) Completed Trial (Per Protocol) with available MRS data: 11 Pts.
Measure: Mean (Standard Deviation); unit: mmol/L, approx. (institutional units)
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 6 | 8
mmol/L, approx. (institutional units)
  Available MRS Secondary Outcomes | 0.7855 (0.8485) | 0.4759 (0.8174)
  Completed Trial (Per Protocol): number analyzed (Participants) | 4 | 7
  Completed Trial (Per Protocol) | 0.5373 (0.8859) | 0.3022 (0.7404)
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; Comparisons of change from W0 to W24 between treatment and placebo are based on a mixed effects regression model using a two-sided Wald test of the interaction term for treatment and time; Test type: Superiority; p > 0.25, Wald test, two-sided — The threshold for statistical significance was p = 0.05

7. Secondary Outcome: Neuroimaging Markers: SV-MRS, Myoinositol, Frontal White Matter, Week 24 Visit Value Minus Baseline Value
Description: Single voxel-magnetic resonance spectroscopy (SV-MRS) myoinositol in frontal white matter. Results were reported as concentrations measured in approximated mmol/L (institutional units).
Time Frame: Changes between baseline and week 24 visits
Population: MRS was performed at both baseline and 24 Weeks on 16 participants (Pts). However, three Pts had invalid frontal white matter MRS results at either baseline or Week 24, and a fourth is missing all Week 24 MRS results due to technical error in data collection.
  Available MRS (data for outcome measure): 12 Pts. (Note: one of the Pts did not complete trial, two were Intent-to-Treat) Completed Trial (Per Protocol) with available MRS data: 9 Pts
Measure: Mean (Standard Deviation); unit: mmol/L, approx. (institutional units)
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 6 | 6
mmol/L, approx. (institutional units)
  Available MRS Secondary Outcomes | 0.2617 (1.8493) | 0.2155 (1.1215)
  Completed Trial (Per Protocol): number analyzed (Participants) | 4 | 5
  Completed Trial (Per Protocol) | 0.6063 (2.1711) | 0.0382 (1.1560)
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p > 0.25, Wald test, two-sided; The threshold for statistical significance was p = 0.05

8. Secondary Outcome: Neuroimaging Markers: SV-MRS, Choline, Basal Ganglia, Week 24 Visit Value Minus Baseline Value
Description: Single voxel-magnetic resonance spectroscopy (SV-MRS) choline in basal ganglia. Results were reported as concentrations measured in approximated mmol/L (institutional units).
Time Frame: Changes between baseline and week 24 visits
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L, approx. (institutional units)
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 6 | 8
mmol/L, approx. (institutional units)
  Available MRS Secondary Outcomes | -0.1495 (0.3583) | 0.1907 (0.4769)
  Completed Trial (Per Protocol): number analyzed (Participants) | 4 | 7
  Completed Trial (Per Protocol) | -0.1905 (0.4548) | 0.1162 (0.4757)
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.244, Wald test, two-sided; Unstandardized beta coefficient = -0.32, Standard Error of Mean 0.27

9. Secondary Outcome: Neuroimaging Markers: SV-MRS, Choline, Frontal White Matter, Week 24 Visit Value Minus Baseline Value
Description: Single voxel-magnetic resonance spectroscopy (SV-MRS) choline in frontal white matter. Results were reported as concentrations measured in approximated mmol/L (institutional units).
Time Frame: Changes between baseline and week 24 visits
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L, approx. (institutional units)
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 6 | 6
mmol/L, approx. (institutional units)
  Available MRS Secondary Outcomes | 0.1670 (0.3430) | -0.1557 (0.2130)
  Completed Trial (Per Protocol): number analyzed (Participants) | 4 | 5
  Completed Trial (Per Protocol) | 0.2028 (0.4017) | -0.2128 (0.1795)
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p > 0.25, Wald test, two-sided — The threshold for statistical significance was p = 0.05

10. Secondary Outcome: Neuroimaging Markers: SV-MRS, N-acetyl Aspartate, Basal Ganglia, Week 24 Visit Value Minus Baseline Value
Description: Single voxel-magnetic resonance spectroscopy (SV-MRS) N-acetyl aspartate concentrations in basal ganglia. Results were reported as concentrations measured in approximated mmol/L (institutional units).
Time Frame: Changes between baseline and week 24 visits
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L, approx. (institutional units)
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 6 | 8
mmol/L, approx. (institutional units)
  Available MRS Secondary Outcomes | -0.5572 (0.9270) | -0.1870 (0.8497)
  Completed Trial (Per Protocol): number analyzed (Participants) | 4 | 7
  Completed Trial (Per Protocol) | -0.7895 (1.1018) | -0.2915 (0.8801)
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p > 0.25, Wald test, two-sided; The threshold for statistical significance was p = 0.05

11. Secondary Outcome: Neuroimaging Markers: SV-MRS, N-acetyl Aspartate, Frontal White Matter, Week 24 Visit Value Minus Baseline Value
Description: Single voxel-magnetic resonance spectroscopy (SV-MRS) N-acetyl aspartate concentrations in frontal white matter. Results were reported as concentrations measured in approximated mmol/L (institutional units).
Time Frame: Changes between baseline and week 24 visits
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L, approx. (institutional units)
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 6 | 6
mmol/L, approx. (institutional units)
  Available MRS Secondary Outcomes | 0.1050 (1.7154) | 0.1432 (0.6497)
  Completed Trial (Per Protocol): number analyzed (Participants) | 4 | 5
  Completed Trial (Per Protocol) | 0.2597 (2.1606) | 0.1134 (0.7218)
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p > 0.25, Wald test, two-sided; The threshold for statistical significance was p = 0.05

12. Secondary Outcome: Neuroimaging Markers: DTI, Whole Brain Mean Fractional Anisotropy (FA), Week 24 Visit Value Minus Baseline Value
Description: Diffusion tensor imaging (DTI), change in whole brain fractional anisotropy (FA) between baseline and 24 weeks. FA is a unitless index that is used for measuring diffusion asymmetry. FA values range from 0 to 1 (0 equals no anisotropy; greater anisotropy is indicated by higher FA values approaching the maximum of 1). FA was measured in regions of interest (ROI) automatically generated by the multi-atlas label-fusion method implemented in the MRICloud. Whole brain mean FA = (Sum of (each ROI's FA * volume)) / (Sum of all ROI volumes).
Time Frame: Changes between baseline and week 24 visits
Population: MRS was performed at both baseline and 24 Weeks on 16 participants (Pts). However, one is missing all Week 24 DTI results due to technical error in data collection.
  Available MRS (data for outcome measure): 15 Pts. (Note: one of the Pts did not complete trial, two were Intent-to-Treat) Completed Trial (Per Protocol) with available MRS data: 12 Pts
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 7 | 8
index
  All Available | -0.0011885 (0.0055178) | -0.0043236 (0.0071927)
  Per Protocol: number analyzed (Participants) | 5 | 7
  Per Protocol | -0.0022483 (0.0035673) | -0.0048070 (0.0076274)
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; Analysis for All Available group (participants who had both Baseline and Week 24 scans); Test type: Superiority; p = 0.366, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees of freedom = 13; Mean Difference (Net) = 0.0031351
Statistical Analysis 2: Comparison: Insulin, Intranasal vs Placebo, Intranasal; Analysis for Per Protocol group; Test type: Superiority; p = 0.505, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees fo freedom = 10; Mean Difference (Net) = 0.0025586

13. Secondary Outcome: Neuroimaging Markers: Diffusion Weighted Imaging, Whole Brain Mean Diffusivity, Week 24 Visit Value Minus Baseline Value
Description: Diffusion weighted imaging, change in whole brain mean diffusivity (MD) between baseline and 24 weeks. MD was measured as the mean of three eigenvalues and has the unit m^2/s. Higher values indicate greater diffusivity. MD was measured in regions of interest (ROI) automatically generated by the multi-atlas label-fusion method implemented in the MRICloud. Whole brain mean MD = (Sum of (each ROI's MD * volume)) / (Sum of all ROI volumes).
Time Frame: Changes between baseline and week 24 visits
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: m^2/s
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 7 | 8
m^2/s
  All Available | 4.7274*10^-6 (1.9275*10^-5) | 4.1177*10^-6 (6.2060*10^-5)
  Per Protocol: number analyzed (Participants) | 5 | 7
  Per Protocol | 5.8845*10^-6 (2.2223*10^-5) | 1.1278*10^-5 (6.3362*10^-5)
Statistical Analysis 1: Comparison: Insulin, Intranasal vs Placebo, Intranasal; Analysis for All Available group (participants who had both Baseline and Week 24 scans); Test type: Superiority; p = 0.98, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees of freedom = 13; Mean Difference (Net) = 0.00000061
Statistical Analysis 2: Comparison: Insulin, Intranasal vs Placebo, Intranasal; Analysis for Per Protocol group; Test type: Superiority; p = 0.86, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Degrees of freedom = 10; Mean Difference (Net) = -0.0000054

14. Secondary Outcome: Neuroimaging Markers: ASL, Week 24 Visit Value Minus Baseline Value
Description: Arterial spin labeling (ASL), a novel measure of cerebral blood flow
Time Frame: Changes between baseline and week 24 visits
Population: Collected data were not considered valid due to an equipment malfunction.
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were reported monthly over the 24-week period that each participant was on study or when taken off study if he/she did not complete the trial. Participants who completed the trial were followed up to 4 weeks after taking the last dose of the investigational product. Participants who stopped the intervention early remained on study for continued follow-up, to the extent possible, through study visits, telephone communication, and medical record review for intent-to-treat analysis.
Arm/Group | Insulin, Intranasal | Placebo, Intranasal
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/11
Other Adverse Events (participants affected / at risk) | 10/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin, Intranasal (N=10) | Placebo, Intranasal (N=11)
Major depressive episode (Psychiatric disorders) | 0 (0) | 2 (2)
Kidney obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Cardiac event (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization for syncope/hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin, Intranasal (N=10) | Placebo, Intranasal (N=11)
Fall (General disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Nosebleed (General disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Congestion/Runny Nose (General disorders) | 4 (4) | 3 (3)
Nasal Irritation or Reaction (during administration of investigational product) (General disorders) | 7 (7) | 4 (4)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Odor/Taste (during administration of investigational product) (Product Issues) | 5 (5) | 1 (1)
Accidental Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Upper Gastrointestinal Pain or Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infection (other than upper respiratory infection) (Infections and infestations) | 2 (2) | 0 (0)
Creatinine, High Blood (Renal and urinary disorders) | 2 (2) | 2 (2)
Nausea (General disorders) | 3 (3) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Blood Pressure, High (acute) (General disorders) | 0 (0) | 1 (1)
Edema, Lower Extremity (General disorders) | 0 (0) | 1 (1)
Glucose, High Blood (Endocrine disorders) | 1 (1) | 0 (0)
Amylase, High Blood (Endocrine disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT03081117/Prot_SAP_001.pdf